CLINICAL TRIAL: NCT02108756
Title: Efficacy and Safety of L-Pantoprazole Sodium Injection to Treat Upper Gastrointestinal Ulcer Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-CTTQ-SPAN
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Bleeding Gastric Ulcer; Bleeding Duodenal Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-pantoprazole sodium (Experimental)
  Interventions: Drug: L-pantoprazole sodium
- Panmeilu (Active Comparator)
  Interventions: Drug: Panmeilu

INTERVENTIONS:
Drug: L-pantoprazole sodium — 2 injection L-pantoprazole sodium (40mg), Bid
  Arms: L-pantoprazole sodium
Drug: Panmeilu — An injection Panmeilu (80 mg) + 1 branch placebo, Bid;
  Arms: Panmeilu

SUMMARY:
The purpose of this study is to evaluate the safety and Efficacy of L- Pantoprazole sodium to treat upper gastrointestinal ulcer bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years, gender:both.
2. Patients whose Forrest classification were in Ⅰ b-Ⅱ c were diagnosed with non-variceal duodenal and / or gastric ulcer bleeding by endoscopy within 24 hours and patients manifested vomiting and / or black stools and other symptoms of upper gastrointestinal bleeding.
3. Patients were diagnosed with upper gastrointestinal bleeding mild to moderate;
4. Informed consent granted.
5. Patients agreed to take medicine and assess.

Exclusion Criteria:

1. Patients were diagnosed with upper gastrointestinal bleeding by endoscopy caused by esophageal varices and portal hypertensive gastropathy, Mallory-Weiss syndrome, dieulafoy disease.
2. Pregnant women or breastfeeding women.
3. Patients who had undergone surgery because of ulcer complications or gastrectomy, gastrointestinal anastomosis within 30 days before the trial.
4. Patients were diagnosed with gastrinoma or gastric malignancy.
5. Patients had other associated complications, which may affect the efficacy.
6. Patients who like alcohol abuse, drug addicts or others which are not suitable for drug trials.
7. Patients who were allergic to any ingredient of any PPI and allergies.
8. Patients diagnosed with small vessel spurting who had to undergo endoscopic hemostasis or surgery or severe gastrointestinal bleeding.
9. Patients suffering from serious heart, brain, lung, liver, kidney disease or severe hypertension.
10. Patients who had coagulopathy, whose PT wasmore three seconds than normal controls, whose APTT> 1.5 times the upper limit of normal or low-dose heparin treatment.
11. Patients whose systolic blood pressure less than 90mmHg or lower > 30mmHg than the baseline systolic blood pressure, pulse pressure less than 20mmHg, hematocrit less than 20%.
12. Patients who participated in other clinical trials within three months before this trial.
13. Patients who need to use other drugs which may affect the trial during the trial or a week before the trial.
14. Patients who were considered unsuitable for selected candidates.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Hemostatic success rate | 6 days

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of the Fourth Military Medical University, Xi'an, Shaanxi, China